CLINICAL TRIAL: NCT02923830
Title: Maintaining Patency in BioFlo Implanted Port Catheters With Saline Only Flushes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We stopped inserting BioFlo ports, no more patients to recruit
Sponsor: TriHealth Inc. (Other)
Responsible Party: Principal Investigator, Rachel Baker, Nurse Researcher, TriHealth Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-117
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Obstruction; Catheter, Infusion Catheter (Vascular); Catheter; Complications (Indwelling Catheter)
MeSH Terms: conditions — Bites and Stings | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Heparinized saline catheter flush - The control group will have their port catheters flushed with 20mL saline + 5mL heparin 100 units/mL; q 3 months
  Interventions: Other: Heparinized saline catheter flush
- Intervention Group (Experimental): Saline-only catheter flush - The intervention group will have their port catheters flushed with saline only.
  Interventions: Drug: Saline-only catheter flush

INTERVENTIONS:
Other: Heparinized saline catheter flush — The control group will have their port catheters flushed with 20mL saline + 5mL heparin 100 units/mL; q 3 months
  Other Names: Control group
  Arms: Control Group
Drug: Saline-only catheter flush — The intervention group will have their port catheters flushed with saline only.
  Other Names: Intervention group
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to determine the safest and most effective flushing solution for maintaining patency (unobstructed flow) in BioFlo implanted port catheters. The complication rate in patients whose ports are flushed with saline only will be compared to the complication rate in patients whose ports are flushed with a combination of saline and heparinized saline.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safest and most effective flushing solution for maintaining patency (unobstructed flow) in BioFlo implanted port catheters. The complication rate in patients whose ports are flushed with saline only will be compared to the complication rate in patients whose ports are flushed with a combination of saline and heparinized saline. These complications include partial or complete obstruction, infection of the central line, and/or the onset of heparin induced thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand English
* Has a BioFlo implanted port in place less than one (1) year
* Evidence of a patent BioFlo port catheter prior to enrollment in the study
* Is receiving active treatment (i.e., receiving a therapeutic drug) through the BioFlo implanted port
* Current treatment protocol projected to continue for a minimum of three (3) months
* Anticipates receiving care at the identified centers for 12 months following enrollment in the study
* Does not receive care of BioFlo implanted port at any other facility

Exclusion Criteria:

* Has documented heparin platelet antibody (i.e., could not be randomized to either group) or other allergy to heparin
* Receiving therapeutic dose of an anticoagulant (e.g.,warfarin, heparin, enoxaparin)
* Does not meet one or more of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Sanker, RN, OCN, Principal Investigator — TriHealth Cancer Institute
Locations (6):
- United States (6):
  - TriHealth Cancer Institute Good Samaritan Infusion Center at GSH, Cincinnati, Ohio
  - Ambulatory Treatment Center at Bethesda North TriHealth Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute Good Samaritan Infusion Center, Medicenter, Cincinnati, Ohio
  - TriHealth Cancer Institute Good Samaritan Infusion Center, Cheviot, Cincinnati, Ohio
  - TriHealth Cancer Institute Good Samaritan Infusion Center, Anderson, Cincinnati, Ohio
  - TriHealth Cancer Institute Good Samaritan Infusion Center Butler County, Hamilton, Ohio

IPD SHARING:
Plan to Share IPD: No
Study terminated

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 13 | 15
Completed | 0 (Study terminated) | 0 (Study terminated)
Not Completed | 13 | 15
Not completed — Physician Decision | 13 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 13 | 20
  >=65 years | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.67 (16.72) | 53.87 (15.20) | 57.78 (16.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 15 | 28
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Occurrence of First Complete Occlusion (Blockage)
Description: Number of Participants with Occurrence of First Complete Occlusion (Blockage) over the 1 year. The date of the first complete occlusion will be recorded.
Time Frame: baseline to 1 year
Population: Study was closed before enrolled subjects completed 12 months of data collection. Data were not analyzed.
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Participants With Occurrence of First Partial Occlusion (Blockage)
Description: Number of Participants with Occurrence of First Partial Occlusion (Blockage) within the 1 year. The date of the first partial occlusion will be recorded.
Time Frame: baseline to 1 year
Population: Study was closed before enrolled subjects completed 12 months of data collection. Data were not analyzed.
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Participants Who Required CathFlo (Alteplase) to Resolve an Occlusion
Description: Number of Participants who required CathFlo (alteplase) to resolve an Occlusion over the 1 year. The date of first CathFlo administration will be recorded.
Time Frame: baseline to 1 year
Population: Study was closed before enrolled subjects completed 12 months of data collection. Data were not analyzed.
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Complete or Partial Occlusions
Description: The number of complete or partial occlusions after the first occurrence will be recorded.
Time Frame: baseline to 1 year
Population: Study was closed before enrolled subjects completed 12 months of data collection. Data were not analyzed.
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Days Catheter Remains Patent (Unobstructed)
Description: The number of days from study enrollment to the first partial or complete occlusion and the number of days between incidences of partial or complete occlusion will be recorded.
Time Frame: baseline to 1 year
Population: Study was closed before enrolled subjects completed 12 months of data collection. Data were not analyzed.
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Central Line-Associated Blood Stream Infection (CLABSI)
Description: Any laboratory-confirmed blood stream infection that is considered central line associated will be recorded.
Time Frame: baseline to 1 year
Population: Study was closed before enrolled subjects completed 12 months of data collection. Data were not analyzed.
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Heparin-related Complication
Description: Heparin Induced Thrombocytopenia (HIT) as measured by a positive HIT antibody test, or any other heparin allergy, will be recorded.
Time Frame: baseline to 1 year
Population: Study was closed before enrolled subjects completed 12 months of data collection. Data were not analyzed.
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 13 months
Description: Plan was to report adverse events to IRB and discuss at study team meeting monthly.
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT02923830/Prot_SAP_000.pdf